CLINICAL TRIAL: NCT04240964
Title: Studying on the Difference Between Foot Osteomyelitis Patients With or Without Diabetes
Brief Title: Studying on the Difference Between Two Kinds of Osteomyelitis
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Ying Cao, associate professor, Nanfang Hospital, Southern Medical University
Other Study IDs: NFEC-2017-013
Record Dates: First submitted 2019-10-28; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Diabetic Foot Osteomyelitis; Diabetic Foot Infection; Microbiome
Keywords: Diabetic Foot Osteomyelitis; 16S rRNA; Metagenomes; Microbiome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dd group: Patients with diabetic foot osteomyelitis
- ND group: Foot osteomyelitis without diabetes

INTERVENTIONS:
Other:

SUMMARY:
To explore the microbial differences of diabetic foot osteomyelitis and osteomyelitis without diabetes.

DETAILED DESCRIPTION:
Diabetic foot osteomyelitis (Dd group) subjects (sample size ≥ 10 cases) and foot osteomyelitis without diabetes (ND group) subjects (sample size ≥ 10 cases) were collected in accordance with the inclusion criteria. Surgeons collected intra-operative bone specimens from all 28 patients who required surgical intervention (debridement or amputation) for management of their osteomyelitis[10]. Avoided soft tissue or sinus tract cultures, because they were not sufficiently accurate in predicting bone pathogens[11]. Following surgical debridement of infected or necrotic tissue, cleansed by sterile saline solution, deep bone specimens were harvested using sterile instruments. We routinely obtained adequate bone specimens and divided them into three parts. One for routine microbiology culture and antibiotic sensitivity testing, one for the histopathology, and the other one for DNA sequencing analysis. This process to obtain bone specimens could reduce chances of contamination by wound tissue colonizing bacteria.

16S rRNA high-throughput sequencing Two specimens were sent to the laboratory for conventional culturing and histopathological tests. The bone specimen left were placed in sterile pipes without any transport medium and stored at 4℃ for 24 hours and then frozen at -80C until DNA extraction. Genomic DNA was extracted using DNA extraction kit (YiRui,ShenZhen,China) according to the manufacturer's instructions. Extracted DNA was quantitative and quality control by agarose gel electrophoresis(JS-power 300, PeiQin, ShangHai, China). Then we amplified the V3-V4 variable region of the 16S rRNA gene for sequencing using a forward and a reverse fusion primer-（341F：5'-CCTAYGGGRBGCASCAG-3' and 806R：5'-GGACTACNNGGGTATCTAAT-3）(ABI GeneAmp 9700 PCR Instrument). PCR products were amplified by removing short sequences, singleton sequences and noisy reads. The PCR reaction was performed in a total volume of 60 μl, containing 6 μl of 10× Ex Tap PCR buffer, 6 μl of dNTP mixture, 0.6μl of bovine serum albumin (BSA), 0.3 μl Ex Tag, 1μl DNA, 1.2μl forward and reverse primers, and 43.7 μlH 2O. The PCR amplification was conducted under following conditions: initial denaturing was conducted at 94°Cfor5min, which was followed by 27 cycles at94°Cfor30s, 55°Cfor30s, and72°C for 45s. A final extension was performed at 72°C for 10min from 28 samples (including DFO and SFO patients) were sequenced over two separate runs on Illumina Miseq. To get high-quality clean reads, raw reads were filtered according to the following rules: (1) remove reads containing morethan10% ofunknown nucleotides and(2) removereads containing less than 80% of bases with quality (Q-value)>20. The filtered reads were then assembled into tags according to overlap between paired-end reads with more than 10bp overlap, and less than 2% mismatch. The software Mothur (v.1.34.0) was used to remove the redundant tags to get unique tags. The obtained unique tags were then used to calculate the abundance.Then we clustered sequences into operational taxonomic units (OTUs) using the Greengene. Taxonomy was assigned to OTUs using the BLASTto the Greengene database at 97% similarity to identify microorganisms at the genera level (species level where possible). A phylogenetic tree was built from aligned representative OTU sequences using figtree.The total species diversity in a landscape was determined by two different parameters, the mean species diversity in sites or habitats at a more local scale (alpha diversity) and the differentiation among those habitats (beta diversity). Alpha diversity included both community diversity and richness: community richness was represented by the ACE estimator or the Chao1 estimator. Beta diversity was the calculation of differences(distance) between microbiome community structure and membership based on the evolution of species. This kind of distance was calculated using Weighted Unifrac and can be performanced by Principal Co-ordinates Analysis diagram.

Metagenomes Analysis A metagenome DNA libraries from specimens were constructed using TruSeq Nano DNA kit (FC-121-4002) according to the manufacturer's instructions, with slight modifications. In brief, the length conformed DNA(350 bp) was obtained by sonication. DNA fragments were end-repaired and the appropriate library size was selected, then the samples were A-tailed and ligated to adapters. The NovaSeq 6000 sequencing systems（Illumina）were used for sequencing and library validation Raw Data obtained by sequencing have a certain proportion of low-quality dataaccording to the following rules: (1) remove reads containing morethan10% ofunknown nucleotides and(2) removereads containing less than 80% of bases with quality (Q-value)>20 . Megahit was used to splice the sequences（clean data） after quality control, and contigs were obtained.Contigs were filtered below 1000bp. The vector and host sequences were filtered by BLASTN, with an E-value cutoff of 1e-5. The remaining reads were mapped to the human genome by SOAP alignment, and the matching reads were removed as being contaminants from the host genome.The taxonomic classifications were performed on assembled contigs and singletons using BLAST against the NCBI database. And the best BLAST hit was used to refer the taxonomic rank of each sequence. All the analyses have been performed in R and p values were corrected for multiple testing with the false discovery rate method.

ELIGIBILITY:
Inclusion Criteria:

1. age≥18 years old.
2. diagnosed as foot osteomyelitis, and wounds were located below the knee joint.
3. nfected bone exposure or positive probe-to-bone test.
4. The patients were good physical condition.
5. Patients were able to tolerate debridement or operation treatment.
6. patients and their families agreed to participate in the study.

Exclusion Criteria:

1. Serious skin diseases around the wound surface;
2. tumors affecting the wound of osteomyelitis;
3. long-term use of immunosuppressive therapy before admission;
4. patients that do not cooperate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with osteomyelitis
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Composition and Diversity of DFO with 16S rRNA Gene Data | 2017-2018
  Subjects who met the inclusion criteria for diabetic foot osteomyelitis (DFO) (sample size ≥ 10) and osteomyelitis without NDFO (sample size ≥ 10) were collected for debridement and amputation for 16s rDNA high-throughput sequencing. Compare microbe composition and diversity between the two groups.
Composition of the DFO Metagenome | 2018-2019
  Subjects who met the inclusion criteria for diabetic foot osteomyelitis (DFO) (sample size ≥ 10) and osteomyelitis without NDFO (sample size ≥ 10) were collected for debridement and amputation for Metagenomic Analysis. Compare microbe composition and diversity between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: ying cao, doctor, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Endocrinology and Metabolism, NanFang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lavery LA, Peters EJ, Armstrong DG, Wendel CS, Murdoch DP, Lipsky BA. Risk factors for developing osteomyelitis in patients with diabetic foot wounds. Diabetes Res Clin Pract. 2009 Mar;83(3):347-52. doi: 10.1016/j.diabres.2008.11.030. Epub 2008 Dec 30. PMID 19117631
- [Background] Berendt AR, Peters EJ, Bakker K, Embil JM, Eneroth M, Hinchliffe RJ, Jeffcoate WJ, Lipsky BA, Senneville E, Teh J, Valk GD. Diabetic foot osteomyelitis: a progress report on diagnosis and a systematic review of treatment. Diabetes Metab Res Rev. 2008 May-Jun;24 Suppl 1:S145-61. doi: 10.1002/dmrr.836. PMID 18442163
- [Background] Valabhji J, Oliver N, Samarasinghe D, Mali T, Gibbs RG, Gedroyc WM. Conservative management of diabetic forefoot ulceration complicated by underlying osteomyelitis: the benefits of magnetic resonance imaging. Diabet Med. 2009 Nov;26(11):1127-34. doi: 10.1111/j.1464-5491.2009.02828.x. PMID 19929991
- [Background] Huang Y, Cao Y, Zou M, Luo X, Jiang Y, Xue Y, Gao F. A Comparison of Tissue versus Swab Culturing of Infected Diabetic Foot Wounds. Int J Endocrinol. 2016;2016:8198714. doi: 10.1155/2016/8198714. Epub 2016 Mar 30. PMID 27123004
- [Background] Goda A, Maruyama F, Michi Y, Nakagawa I, Harada K. Analysis of the factors affecting the formation of the microbiome associated with chronic osteomyelitis of the jaw. Clin Microbiol Infect. 2014 May;20(5):O309-17. doi: 10.1111/1469-0691.12400. Epub 2013 Nov 11. PMID 24112138
- [Background] Redel H, Gao Z, Li H, Alekseyenko AV, Zhou Y, Perez-Perez GI, Weinstock G, Sodergren E, Blaser MJ. Quantitation and composition of cutaneous microbiota in diabetic and nondiabetic men. J Infect Dis. 2013 Apr;207(7):1105-14. doi: 10.1093/infdis/jit005. Epub 2013 Jan 8. PMID 23300163
- [Derived] Zou M, Cai Y, Hu P, Cao Y, Luo X, Fan X, Zhang B, Wu X, Jiang N, Lin Q, Zhou H, Xue Y, Gao F. Analysis of the Composition and Functions of the Microbiome in Diabetic Foot Osteomyelitis Based on 16S rRNA and Metagenome Sequencing Technology. Diabetes. 2020 Nov;69(11):2423-2439. doi: 10.2337/db20-0503. Epub 2020 Aug 14. PMID 32801139